CLINICAL TRIAL: NCT02344459
Title: Randomized Controlled Trial: Comparing 30mL Single Versus 80mL Double Balloon Catheters for Pre-induction Cervical Ripening
Brief Title: Comparing 30mL Single Versus 80mL Double Balloon Catheters for Pre-induction Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kara Hoppe, Maternal Fetal Medicine Fellow, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36685-D
Record Dates: First submitted 2014-12-01; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Pre-induction Cervical Ripening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 80mL double balloon catheter (Cook catheter®) (Experimental)
  Interventions: Device: mechanical pre-induction cervical ripening
- 30mL single Foley balloon catheter (Active Comparator)
  Interventions: Device: mechanical pre-induction cervical ripening

INTERVENTIONS:
Device: mechanical pre-induction cervical ripening — The balloon catheters have been used to provide mechanical dilation to the cervix as a method of pre-induction cervical ripening.

SUMMARY:
The purpose of this study is to perform a randomized controlled trial to compare the efficacy of 80mL double balloon catheter versus a 30mL single catheter balloon for pre-induction cervical ripening by evaluating the change in Bishop score.

ELIGIBILITY:
Inclusion Criteria:

* Bishop score of 5 or less
* Singleton
* Cephalic presentation
* Fewer than 4 contractions in 10 minutes
* Reactive fetal monitoring

Exclusion Criteria:

* Non-vertex presentation
* Placenta previa
* Vasa previa
* Unexplained vaginal bleeding
* Active herpes simplex virus infection
* Non-English speaking
* Previous attempt at an induction of labor in the current pregnancy
* Prolapsed umbilical cord
* More than one prior cesarean delivery or history of classical cesarean delivery
* Patients receiving or planning to undergo exogenous prostaglandin administration as the primary induction agent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bishop score greater than or equal to 6 at time of balloon catheter removal | until catheter removal (12 hours maximum)

SECONDARY OUTCOMES:
induction to delivery time | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
vaginal delivery time less than 24 hours from initiation of induction | 24 hours
mode of delivery | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
Time to catheter expulsion | Up to 12 hours
Type of catheter expulsion | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
  spontaneous vs. provider
Epidural utilization | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
Meconium stained amniotic fluid | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
5 minute Apgar score | The participants infant will be monitored from immediately to 5 minutes after birth
Medication required to augment labor | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
  prostaglandins, oxytocin
Artificial rupture of membranes required to augment labor | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
Cesarean section indications | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
Neonatal intensive care unit admissions | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
Chorioamnionitis | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)
birthweight | The participant will be monitored from time of admission until delivery, an expected average of 24-48 hours of the infant (on average 24-48 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Kara K Hoppe, DO, Principal Investigator — University of Washington